CLINICAL TRIAL: NCT01241721
Title: Clinical Value of Pre-Surgery Positron Emission Mammography (PEM) in Patients With Newly Diagnosed Breast Cancer
Brief Title: Pre-Surgery Positron Emission Mammography in Patients With Newly Diagnosed Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRC 09096
Record Dates: First submitted 2010-10-06; First posted 2010-11-16 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer; Breast Cancer Surgery
Keywords: Breast Diseases; Breast Neoplasms; Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positron Emission Mammography (PEM) (Experimental): Positron Emission Mammography (PEM)
  Interventions: Device: Positron Emission Mammography (PEM)

INTERVENTIONS:
Device: Positron Emission Mammography (PEM) — Phase 1 of the study will involve imaging the breast with cancer up to 3 times over 2 hours using one half (1/2) of the standard dose of the radioactive tracer, F18FDG, for PEM imaging. If this reduced dose is equivalent to the standard dose then one quarter (1/4) dose will be tested to find the lowest effective radiation dose of tracer to see breast cancer. Phase 2 of the study will involve imaging of both breasts several times over a shorter duration using the lowest effective dose of tracer identified in the first part of the study. This will allow us to examine the reliability of PEM to identify a second unsuspected abnormality in either breast. Patients will be offered biopsy by ultrasound, MRI or PEM as clinically appropriate of lesions suspected of being cancer prior to final surgical planning.

SUMMARY:
The purpose of the study is to determine the optimal, lowest dose of radioactive tracer required for Positron Emission Mammography (PEM), and the accuracy and reliability of PEM in pre-surgical evaluations for patients with newly diagnosed breast cancer anticipating breast-conserving surgery but identified to have a second unsuspected breast cancer by MRI.

DETAILED DESCRIPTION:
The purpose of this research in Phase 1 is to determine the lowest dose of radionuclide 18F-FDG that can be used in the Diagnostic use of Positron Emission Mammography for the diagnosis of multifocal breast cancer in patients wishing to have Breast Conservation Surgery for newly diagnosed breast cancer. Low dose injections (radioactive counts) of 18F-FDG will be compared to the equivalent radioactive counts for the standard higher dose 10 millicuries used in standard PEM studies in current clinical practice. Images will be post processed by computer aided software and will be placed in two categories: Low dose group, and higher dose group. Images will be randomly blinded to readers to assess the ability to see positive lesions that warrant further biopsy or to include in current surgical planning prior to breast conservation surgery or mastectomy. Images will be assessed for ability to see the PEM positive lesions on the lower dose images and this will be compared to the ability to see the PEM positive lesions on the standard higher dose images. Each of three breast cancer categories will be assessed Infiltrating Ductal Carcinoma, Lobular infiltrating Carcinoma, and Ductal Carcinoma Insitu. Phase 1 will have 30 patients.

The purpose of the research in Phase 2 is to use the lowest dose identified in Phase 1 for imaging primary breast cancer patients who have been identified by breast MRI to have an unsuspected second lesion of the breast not expected from Mammography or Ultrasound that requires biopsy for diagnosis prior to the biopsy to compare the reliability of PEM and MRI for identifying breast cancer at the 2nd site. Parameters assessed will include standard statistical analysis for sensitivity, specificity, positive predictive value and negative predictive value for MRI and PEM imaging with the new lower radionuclide dose selected by Phase 1. Phase 2 will have 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Newly diagnosed primary breast cancer
* Must have a breast or breast/chest MRI ordered as part of standard of care
* Must meet one or more of the following in Part 1:

  * T1 carcinoma of the breast appropriate for breast conserving surgery diagnosis established by core biopsy
  * Tis (ductal carcinoma in situ) carcinoma > 2 cm diameter
  * Invasive lobular carcinoma of the breast
* Must meet the following in Part 2:

  * Known invasive or in situ primary breast cancer identified on pre-surgical breast MRI to have an unsuspected 2nd lesion recommended for biopsy and biopsy has not yet been performed

Exclusion Criteria:

* Known diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
PEM identification of primary breast cancer. | Upon study completion (~3 years)

SECONDARY OUTCOMES:
Lowest dose of F18-FDG giving optimal PEM imaging of primary breast cancers. | After the first 30 subjects (~one year)
Identification of 2nd unsuspected primary breast cancer by PEM in patients with known index primary breast cancer. | Upon study completion (~3 years)
Comparison of PEM and MRI for identification of index primary breast cancer and unsuspected primary breast cancer. | Upon study completion (~3 years)
Comparison of PEM and MRI for identification of breast lesions that require biopsy but are not an unsuspected 2nd primary breast cancer in patients with known index primary breast cancer. | Upon study completion (~3 years)

CONTACTS AND LOCATIONS:
Overall Officials: J. David Beatty, MD, Principal Investigator — Swedish Medical Center Cancer Institute
Locations (2):
- United States (2):
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Cancer Institute Cherry Hill Campus - Comprehensive Breast Center, Seattle, Washington